CLINICAL TRIAL: NCT03397108
Title: Assessing the Drug Exposure Risk of Infants Breastfed by Women With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Shinya Ito, Principal Investigator, Head of Clinical Pharmacology & Toxicology, The Hospital for Sick Children
Other Study IDs: 1000056982
Record Dates: First submitted 2017-12-19; First posted 2018-01-11 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Healthy Controls
Keywords: Inflammatory Bowel Disease; Crohn disease; Colitis; TNF; Breast milk; monoclonal antibody
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Colitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human milk samples will be collected and analyzed for TNF alpha, TNF alpha-dependent chemokines, and infliximab/adalimumab levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with IBD: This group is composed of breastfeeding women aged over 18 years and in their first 4-month postpartum period, who are diagnosed with Crohn's disease or Ulcerative Colitis. Some of them were receiving anti-TNF monoclonal antibody prescribed by their prescribers (outside this observational study) at a standard dose and interval.
  Interventions: Other: The IBD group was divided into 2 subgroups: with or without anti-TNF antibody use
- Healthy breastfeeding women: This group is composed of healthy breastfeeding women aged over 18 years and in their first 4-month postpartum period.

INTERVENTIONS:
Other: The IBD group was divided into 2 subgroups: with or without anti-TNF antibody use — This observational study enrolled women with IBD, and some of them were receiving a treatment with anti-TNF monoclonal antibody, which was prescribed by their responsible prescribers at a standard dose and dosing interval.
  Groups: Women with IBD

SUMMARY:
Breastfeeding is beneficial to both mother and baby. However, many breastfeeding women are affected by long-term health conditions and need to take medications.

Inflammatory Bowel Disease (IBD) is marked by an abnormal response of the body's immune system, and high levels of certain proteins that cause inflammation (Cytokines like Tumor Necrosis Factor-alpha or TNF). A group of drugs called "biologics" target and stop these proteins from causing inflammation, and have been successfully used to treat this condition. Inflammatory proteins may be present in breast milk of healthy women in variable levels, and may play a role in development of infant's brain and immune system.

This observational study is conducted to investigate:

* Concentration of some of the inflammatory proteins in breast milk of mothers with IBD and healthy controls
* Interaction between these proteins and biologics in breast milk of women with IBD
* Potential role of these proteins (and their interaction with biologics) on development of infant learning and memory function It has been presumed that concentrations of TNF and some other cytokines are higher in breast milk of women with IBD, and the biologics can normalize these high levels.

Note: Due to the pandemic, the study now consists of reduced number of study visits. The mandatory visits include two home visits in the first 4 months postpartum to complete a participant questionnaire and collect a small sample of breast milk at each visit. The optional study visits consist of two visits at the Hospital for Sick Children for evaluation of learning and memory function of the infant at the ages of 12 and 18 months. Additionally, mothers will be required to complete for their infant subscales of The Ages and Stages Questionnaires®, Third Edition (ASQ®-3) either in person or over the telephone at the ages of 12 months and 18 months.

DETAILED DESCRIPTION:
The inflammatory bowel disease (IBD) shows the highest incidence among people of childbearing age. Indeed, it is not uncommon that pregnant or lactating women with IBD require drug therapy, including monoclonal antibodies against Tumor Necrosis Factor-alpha (TNF).

TNF and TNF-dependent chemokines are normally expressed in milk. Importantly, experimental data indicate enhanced brain growth and cognitive development in the mouse offspring given milk deficient in TNF and TNF-dependent chemokines. Patients with IBD are often treated with monoclonal antibodies against TNF (TNFmAb). Although TNFmAb is used during breastfeeding due to their minimal milk excretion, whether it affects endogenous TNF/chemokines in human milk is not known.

Our hypotheses are: 1) Women with IBD have higher TNF (and TNF-dependent chemokines) in milk than non-IBD control women, because of the inflammatory condition; and 2) Women with IBD receiving TNFmAb have lower TNF (and TNF-dependent chemokines) in milk than those with IBD who are not treated with TNFmAb.

We conduct an observational study of breastfeeding women with or without IBD. Some of these women with IBD are likely to be receiving TNFmAb. We measure milk concentrations of TNF and TNF-dependent chemokines in early (5-6 weeks postpartum) and mid-lactation period (13-14 weeks postpartum). Also, as an exploratory analysis, we assess their infant's cognitive and language development at 12 month and 18 months using Bayley-III tool.

Note:

Because there was no information at the outset of the study on cytokine profiles in milk of women with inflammatory conditions including IBD, a formal sample size could not be estimated. Although a provisional target was set, the study was designed to continue for the planned study duration as no stopping rule had been defined. Also, our original protocol included a population pharmacokinetic study of TNFmAb in milk. However, due to the pandemic and difficulty in developing the assay method, we were not able to start this part of the project.

ELIGIBILITY:
Inclusion Criteria:

* Breastfeeding women with IBD or healthy breastfeeding women in the first 4-month postpartum period

Exclusion Criteria:

* unable to communicate in English
* Present illness of chronic inflammatory conditions (except IBD)
* Mastitis
* Present acute or chronic infection
* use of a different anti-Tumor Necrosis Factor (TNF) drug within the last 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants are required to live in the Greater Toronto Area. The IBD group will be selected from IBD clinics, while the healthy controls will be selected from the community samples who volunteer to participate.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shinya Ito, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Participant-level data collected during the study will be available for research purposes in a form of de-identified individual data upon reasonable request. Other research documents such as study protocol may be also available. This data sharing activity is contingent upon approval from the institutional research ethics board of the Hospital for Sick Children. An interested party may submit a proposal to the study team up to 36 months following article publication, describing the purpose and methods of data use. Data requestors may need to sign a data transfer agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available from February 2025 to January 2028
Access Criteria: 1. Request deemed reasonable by the study team
  2. No objection from the research ethics board of the Hospital for Sick Children
  3. No objection from the legal department of the Hospital for Sick Children

REFERENCES:
- [Background] Maron JL. The importance of investigating the effects of drug therapy on maternal breast milk composition. Pediatr Res. 2025 May;97(6):1765-1766. doi: 10.1038/s41390-024-03785-1. Epub 2024 Dec 13. No abstract available. PMID 39672826
- [Result] Sepiashvili L, Brydon A, Koroshegyi C, Gold A, Dalvi P, Ghayoori S, Rahman M, Huang V, Maxwell C, Nguyen GC, Ito S. Reduction of tumor necrosis factor (TNF) in milk of women receiving anti-TNF antibody. Pediatr Res. 2025 May;97(6):1935-1942. doi: 10.1038/s41390-024-03672-9. Epub 2024 Nov 1. PMID 39487320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between August 2017 to November 2022
Groups:
- Women With IBD: This group is composed of breastfeeding women aged over 18 years and in their first 4-month postpartum period, who are diagnosed with Crohn's disease or Ulcerative Colitis.
Period: Overall Study
Arm/Group | Women With IBD | Healthy Breastfeeding Women
Started | 46 | 33
Completed | 26 | 31
Not Completed | 20 | 2
Not completed — Lost to Follow-up | 15 | 0
Not completed — Insufficient milk production | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women With IBD | Healthy Breastfeeding Women | Total
Number analyzed (Participants) | 26 | 31 | 57
Age, Continuous [Median (Full Range); unit: years] | 34 [28 to 43] | 34 [25 to 39] | 34 [25 to 43]
Sex/Gender, Customized [Number; unit: participants]
  Female | 26 | 31 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 31 | 57
Maternal Weight [Median (Full Range); unit: kg] | 68 [48 to 102] | 66 [50 to 92] | 67 [48 to 102]
Maternal BMI [Median (Full Range); unit: kg/m^2] | 25 [20 to 35] | 24 [19 to 32] | 24.5 [19 to 35]
Pregnancy period [Median (Full Range); unit: week] | 39 [37 to 41] | 39 [36 to 41] | 39 [36 to 41]
Mode of Delivery [Number; unit: participants]
  Vaginal | 16 | 27 | 43
  C-section | 10 | 4 | 14
Infant Sex: Female [Number; unit: participants] | 15 | 13 | 28
Infant birth weight [Median (Full Range); unit: grams] | 3351 [2410 to 4536] | 3402 [2595 to 4170] | 3376.5 [2410 to 4170]
Smoking during pregnancy [Number; unit: participants] | 0 | 0 | 0
Breastfeeding status [Number; unit: participants]
  Exclusive breastfeeding | 16 | 23 | 39
  Predominant (>80% of time) | 8 | 6 | 14
  Usual (<80% of time) | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Levels of TNF (Tumor Necrosis Factor Alpha) and TNF-dependent Chemokines (MCP1, MIP-1beta and IP10) in Breast Milk of Women With IBD and Healthy Controls by Multiplex Assay
Description: This observational study collected milk samples during the defined study periods: early-lactation and mid-lactation. To capture a temporal profiles of Tumour Necrosis Factor (TNF) and TNF-dependent chemokine levels, we analyzed these 2 sampling periods separately, instead of pooling them per sampling period.
  Multiplex assay was used to measure TNF and TNF-dependent downstream chemokines including MCP-1 (CCL2), MIP-1beta (CCL4) and IP10 (CXCL10) in breast milk of two groups of participants (women with IBD and healthy controls) at two sampling periods (early- and mid-lactation). Our original plan included MCP-3 (CCL7) as well, but an average quantification rate for this chemokine was only 33%, and therefore we excluded MCP-3 from our analyses.
Time Frame: Two points at early-lactation (median 5-6 postpartum weeks) and mid-lactation (median 13-14 postpartum weeks)
Population: Control is non-IBD breastfeeding women. IBD group was divided into 2 subgroups based on the status of their treatment with anti-TNF antibody (TNFmAb). Participants were tested twice: first, during early lactation period and second, later during mid-lactation period. Six women in IBD group could not provide milk samples during the mid-lactation period. MCP-3 (CCL7) detection rate was 33% of all samples and therefore excluded from the analyses.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- IBD Subgroup "On TNFmAb Treatment": Those women in the IBD group were further stratified into two subgroups based on the use of anti-TNF monoclonal antibody (TNFmAb): 1) "on TNFmAb treatment" if they received either infliximab within 8 weeks or adalimumab within 2 weeks of sample collection dates, which are usual dosing intervals of TNFmAb maintenance regimens; 2) otherwise "off TNFmAb treatment".
- IBD Subgroup "Off TNFmAb Treatment": Those women in the IBD group were further stratified into two subgroups based on the use of anti-TNF monoclonal antibody (TNFmAb): 1) "on TNFmAb treatment" if they received either infliximab within 8 weeks or adalimumab within 2 weeks of sample collection dates, which are usual dosing intervals of TNFmAb maintenance regimens; 2) if they were not receiving them during the sampling periods, "off TNFmAb treatment".
Arm/Group | Healthy Breastfeeding Women | Women With IBD | IBD Subgroup "On TNFmAb Treatment" | IBD Subgroup "Off TNFmAb Treatment"
Number analyzed (Participants) | 31 | 26 | 9 | 17
pg/ml
  Early-lactation: TNF | 12.5 [9.6 to 28.5] | 19.8 [5.7 to 34.0] | 7.1 [3.1 to 15.8] | 23.5 [9.8 to 49.3]
  Early-lactation: MCP1 | 1078.0 [398.3 to 3383.0] | 1325.0 [317.9 to 2761.0] | 339.6 [201.2 to 1949.0] | 1352.0 [879.1 to 3694.0]
  Early-lactation:MIP1beta | 13.4 [6.6 to 17.9] | 12.6 [6.0 to 27.5] | 7.1 [2.6 to 13.5] | 17.7 [9.2 to 47.6]
  Early-lactation: IP10 | 3985.0 [1355.0 to 6952.0] | 2302.0 [853.5 to 5429.0] | 898.8 [273.7 to 2014.0] | 3360.0 [1511.0 to 10549.0]
  Mid-lactation: TNF: number analyzed (Participants) | 31 | 20 | 5 | 15
  Mid-lactation: TNF | 11.1 [5.6 to 18.6] | 16.4 [6.5 to 21.5] | 7.3 [3.6 to 14.7] | 18.8 [8.1 to 43.6]
  Mid-lactation: MCP1: number analyzed (Participants) | 31 | 20 | 5 | 15
  Mid-lactation: MCP1 | 513.1 [403.4 to 1802.0] | 679.5 [403.4 to 1802.0] | 305.8 [183.8 to 1753.0] | 693.8 [522.3 to 1981.0]
  Mid-lactation: MIP1beta: number analyzed (Participants) | 31 | 20 | 5 | 15
  Mid-lactation: MIP1beta | 8.2 [3.7 to 16.9] | 16.4 [6.7 to 31.0] | 6.9 [1.0 to 20.6] | 18.1 [7.0 to 35.1]
  Mid-lactation: IP10: number analyzed (Participants) | 31 | 20 | 5 | 15
  Mid-lactation: IP10 | 2041.0 [970.3 to 3681.0] | 1277.0 [748.2 to 2785.0] | 981.9 [578.0 to 1758.0] | 1820.0 [745.4 to 4024.0]
  Early-lactation MCP-3 | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics. | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics. | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics. | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics.
  Mid-lactation MCP-3: number analyzed (Participants) | 31 | 20 | 5 | 15
  Mid-lactation MCP-3 | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics. | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics. | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics. | NA [NA to NA] — 67% of MCP-3 (CCL7) were below quantitation limit and was judged inappropriate to derive sample statistics.
Statistical Analysis 1: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk TNF levels at EARLY LACTATION PERIOD were compared between non-IBD control and women with IBD. Our hypothesis was that women with IBD have higher TNF in milk due to the underlying inflammatory condition (IBD); Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — The a priori threshold of significance was set at 0.05. Not adjusted for multiple comparison
Statistical Analysis 2: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk TNF at the EARLY LACTATION PERIOD was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". We hypothesized that the use of TNFmAb decreases milk TNF. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.024, Kruskal-Wallis
Statistical Analysis 3: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk MCP1 levels (TNF dependent chemokine) at the EARLY LACTATION PERIOD were compared between non-IBD control and IBD group to see if there is a difference; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney) — The a priori threshold of significance was set at 0.05. Not adjusted for multiple comparison
Statistical Analysis 4: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk levels of MIP-1 beta (TNF dependent chemokine) at the EARLY LACTATION PERIOD were compared between non-IBD control and IBD group to see if there is a difference; Test type: Superiority; p = 0.93, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison
Statistical Analysis 5: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk IP10 levels (one of the TNF dependent chemokines) at EARLY LACTATION PERIOD were compared between non-IBD control and IBD group to see if there is a difference; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — The a priori threshold of significance was set at 0.05. Not adjusted for multiple comparison
Statistical Analysis 6: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk levels of TNF-dependent chemokine, MCP1, at the EARLY LACTATION PERIOD was compared among the 3 groups: non-IBD control and the 2 IBD subgroups. We hypothesized that the use of TNFmAb decreases milk TNF and TNF-dependent chemokine including MCP1. Nonparametric comparison of the 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.12, Kruskal-Wallis
Statistical Analysis 7: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk MIP-1beta at the EARLY LACTATION PERIOD was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". We hypothesized that the use of TNFmAb decreases milk TNF and TNF-dependent chemokine including MIP-1beta. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.051, Kruskal-Wallis
Statistical Analysis 8: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk IP10 at the EARLY LACTATION PERIOD was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". We hypothesized that the use of TNFmAb decreases milk TNF and TNF-dependent chemokine including IP10. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.0046, Kruskal-Wallis
Statistical Analysis 9: Comparison: Healthy Breastfeeding Women vs Women With IBD; Comparison of milk TNF level at the MID LACTATION POINT between non-IBD control and IBD group. The same analytical framework as the early lactation, but this is based on data at the mid-lactation point (13-14 postpartum weeks). Our hypothesis is the same as for the early-lactation point; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison
Statistical Analysis 10: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk TNF at MID LACTATION POINT was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". Hypothesis is the same as for the early lactation point. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.11, Kruskal-Wallis
Statistical Analysis 11: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk MCP1 level comparison between non-IBD control and IBD group at the MID LACTATION POINT(13-14 postpartum weeks). Our hypothesis is the same as for the early-lactation point; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison
Statistical Analysis 12: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk MIP-1beta level comparison between non-IBD control and IBD group at the MID LACTATION POINT (13-14 postpartum weeks). Our hypothesis is the same as for the early-lactation point; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison
Statistical Analysis 13: Comparison: Healthy Breastfeeding Women vs Women With IBD; Milk IP10 level comparison between non-IBD control and IBD group at the MID LACTATION POINT (13-14 postpartum weeks). Our hypothesis is the same as for the early-lactation point; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison
Statistical Analysis 14: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk MCP-1 at the MID LACTATION PERIOD was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". The hypothesis is the same as that for the early-lactation period. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.21, Kruskal-Wallis
Statistical Analysis 15: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk MIP-1beta at the MID LACTATION POINT was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". The hypothesis is the same as that for the early-lactation period. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.12, Kruskal-Wallis
Statistical Analysis 16: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Milk IP10 at the MID LACTATION POINT was compared among the 3 groups: non-IBD control, IBD subgroup "On TNFmAb" and IBD subgroup "Off TNFmAb". The same hypothesis as that for the early-lactation period. Nonparametric comparison of 3 groups was done with one-way ANOVA on ranks (Kruskal-Wallis test), followed by multiplicity-adjusted pairwise comparisons with Dunn's test; Test type: Superiority; p = 0.29, Kruskal-Wallis
Statistical Analysis 17: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants at the EARLY LACTATION, we analyzed correlation between milk TNF and chemokine MCP1 to see if they are positively correlated. This is to show supportive evidence for TNF dependency of chemokine MCP1; Test type: Other — Correlation analysis; p < 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.7232, 95% CI 2-sided [0.5647 to 0.8303]
Statistical Analysis 18: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants at the EARLY LACTATION, we analyzed correlation between milk TNF and chemokine MIP-1beta to see if they are positively correlated. This is to show supportive evidence for TNF dependency of chemokine MIP-1beta; Test type: Other — Correlation analysis; p < 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.6835, 95% CI 2-sided [0.5088 to 0.8042]
Statistical Analysis 19: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants at the EARLY LACTATION, we analyzed correlation between milk TNF and chemokine IP10 to see if they are positively correlated. This is to show supportive evidence for TNF dependency of chemokine IP10; Test type: Other — Correlation analysis; p < 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.6316, 95% CI 2-sided [0.4377 to 0.7693]
Statistical Analysis 20: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants at the MID LACTATION POINT, we analyzed correlation between milk TNF and MCP1 to see of they are positively correlated; Test type: Other — Correlation analysis; p < 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.5720, 95% CI 2-sided [0.3445 to 0.7360]
Statistical Analysis 21: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants at the MID LACTATION POINT, we analyzed correlation between milk TNF and MIP-1beta to see of they are positively correlated; Test type: Other — Correlation analysis; p < 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.7564, 95% CI 2-sided [0.6022 to 0.8562]
Statistical Analysis 22: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants at the MID LACTATION POINT, we analyzed correlation between milk TNF and IP10 to see of they are positively correlated; Test type: Other — Correlation analysis; p = 0.0227, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.32, 95% CI 2-sided [0.03869 to 0.5520]
Statistical Analysis 23: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants, we assessed temporal tracking of milk TNF between early and mid-lactation points; Test type: Other — Correlation analysis; p = 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.52, 95% CI 2-sided [0.2727 to 0.6975]
Statistical Analysis 24: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants, we assessed temporal tracking of milk MCP1 between early and mid-lactation points; Test type: Other — Correlation analysis; p = 0.0005, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.4722, 95% CI 2-sided [0.2181 to 0.6664]
Statistical Analysis 25: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants, we assessed temporal tracking of milk MIP-1beta between early and mid-lactation points; Test type: Other — Correlation analysis; p = 0.01, Spearman rank correlation — Not adjusted for multiple comparison; Spearman rank correlation = 0.36, 95% CI 2-sided [0.0802 to 0.5803]
Statistical Analysis 26: Comparison: Healthy Breastfeeding Women vs Women With IBD; Using the pooled data of all participants, we assessed temporal tracking of milk IP10 between early and mid-lactation points; Test type: Other — Correlation analysis; p < 0.0001, Spearman rank correlation — Not adjusted for multiple comparison; Spearman r = 0.66 (95%CI: 0.4670 - 0.7964). Number of XY pairs: 51; Spearman rank correlation = 0.66, 95% CI 2-sided [0.4670 to 0.7964]

2. Secondary Outcome: Scores on Cognitive Subset of Bayley Scales of Infant and Toddler Development- Third Version (Bayley-III) in Infants of Healthy Controls and Women With IBD
Description: We used Bayley Scales of Infant and Toddler development- Third Version (Bayley-III): which is used widely to measure child's cognitive and language development. In this scale, for both cognitive and language scores, minimum standard score is 45 and maximum standard score is 155: Higher standard scores indicates stronger/better performance.
  Children of the participating mothers were tested at the age of 12 months and 18 months. The language assessment is also used for comprehensiveness, but this has been added after the study was started. The test is performed as a single-blinded assessment in a controlled environment at the Hospital for Sick Children by a trained psychometrist supervised by a psychologist.
Time Frame: At the infant age of 12 months and 18 months
Population: Language test was introduced to the project for completeness after the study had started. This created lower sample numbers at the 12 month point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Infants Breastfed by Women With IBD: At 12 months of age 15 infants were eligible for the cognitive assessment after their parent provided informed consent for the test.
  8 of the 15 infants were also tested for the language development.
  At 18 months of age 12 infants were eligible for the cognitive assessment after their parent provided informed consent for the test.
  11 of the 12 infants were also tested for the language development.
- Infants Breastfed by Women Without IBD: At 12 months of age 28 infants were eligible for the cognitive assessment after their parent provided informed consent for the test.
  14 of the 28 infants were also tested for the language development.
  At 18 months of age 16 infants were eligible for the cognitive assessment after their parent provided informed consent for the test.
  All 16 infants were also tested for the language development.
Arm/Group | Infants Breastfed by Women With IBD | Infants Breastfed by Women Without IBD
Number analyzed (Participants) | 15 | 28
score on a scale
  Cognitive at 12 month | 103.0 (7.0) | 107.1 (8.8)
  Language at 12 month: number analyzed (Participants) | 8 | 14
  Language at 12 month | 105.4 (9.7) | 107.7 (8.3)
  Cognitive at 18 month: number analyzed (Participants) | 12 | 16
  Cognitive at 18 month | 108.8 (8.6) | 114.7 (10.8)
  Language at 18 month: number analyzed (Participants) | 11 | 16
  Language at 18 month | 107.0 (15.6) | 105.3 (13)
Statistical Analysis 1: Comparison: Infants Breastfed by Women With IBD vs Infants Breastfed by Women Without IBD; Cognitive development at 12 months of age. Animal data suggested that pups receiving milk with lower TNF and TNF-dependent chemokines showed enhanced cognitive development. Because there was no guiding information in humans regarding milk TNF level differences between women with and without IBD, our main goal was to measure milk TNF levels. The infant cognitive/language assessment, therefore, had to be designed as a pilot and exploratory in nature; Test type: Superiority; p = 0.12, t-test, 2 sided
Statistical Analysis 2: Comparison: Infants Breastfed by Women With IBD vs Infants Breastfed by Women Without IBD; Language development at 12 months of age; Test type: Superiority; p = 0.56, t-test, 2 sided
Statistical Analysis 3: Comparison: Infants Breastfed by Women With IBD vs Infants Breastfed by Women Without IBD; Cognitive development at 18 months of age; Test type: Superiority; p = 0.16, t-test, 2 sided
Statistical Analysis 4: Comparison: Infants Breastfed by Women With IBD vs Infants Breastfed by Women Without IBD; Language development at 18 months of age; Test type: Superiority; p = 0.75, t-test, 2 sided
Statistical Analysis 5: Comparison: Infants Breastfed by Women With IBD vs Infants Breastfed by Women Without IBD; Using pooled data of all participants at the early-lactation sample point, correlation between milk TNF levels and 12 month cognitive development was examined to investigate if they were inversely correlated; Test type: Other — Correlation analysis; p = 0.0853, Spearman rank correlation; Spearman rank correlation = 0.2655, 95% CI 2-sided [-0.047 to 0.5307]
Statistical Analysis 6: Comparison: Infants Breastfed by Women With IBD vs Infants Breastfed by Women Without IBD; Using the pooled data of all participants, correlation analysis between milk TNF at early lactation and 12 month language score was done to see if they were inversely correlated; Test type: Other — Correlation analysis; p = 0.090, Spearman rank correlation; Spearman rank correlation = 0.3705, 95% CI 2-sided [-0.07385 to 0.6921]

3. Other Pre Specified Outcome: Population Pharmacokinetic Study of Anti-TNF Monoclonal Antibody in Milk
Description: Concentrations of anti-TNF monoclonal antibody in milk will be measured once the method is validated. The data will be analyzed using population pharmacokinetic modeling.
Time Frame: 1-2 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Milk Sampling Time Point in the Early Lactation Period
Description: This is the early lactation sampling points: one of the two milk sampling time points (post-partum weeks). The milk samples were analyzed for their TNF and chemokine levels.
Time Frame: postpartum weeks until 10 weeks.
Measure: Median (Inter-Quartile Range); unit: postpartum weeks
Arm/Group | Healthy Breastfeeding Women | Women With IBD | IBD Subgroup "On TNFmAb Treatment" | IBD Subgroup "Off TNFmAb Treatment"
Number analyzed (Participants) | 31 | 26 | 9 | 17
postpartum weeks | 5.3 [4.5 to 7.3] | 5.5 [5.0 to 6.5] | 6.0 [5.0 to 6.9] | 5.4 [4.7 to 6.7]
Statistical Analysis 1: Comparison: Healthy Breastfeeding Women vs Women With IBD; This is to confirm that the 2 groups are not different for their sampling time points in the early lactation period; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparison
Statistical Analysis 2: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Test type: Superiority; p = 0.96, Kruskal-Wallis

5. Other Pre Specified Outcome: Milk Sampling Time Point in the Mid Lactation Period
Description: This is the second milk sampling point corresponding to the mid-lactation period.
Time Frame: postpartum weeks of 10-20 weeks.
Measure: Median (Inter-Quartile Range); unit: postpartum weeks
Arm/Group | Healthy Breastfeeding Women | Women With IBD | IBD Subgroup "On TNFmAb Treatment" | IBD Subgroup "Off TNFmAb Treatment"
Number analyzed (Participants) | 31 | 20 | 5 | 15
postpartum weeks | 13.9 [12.3 to 15.1] | 13.3 [12.3 to 14.2] | 13.2 [11.7 to 13.7] | 13.5 [12.3 to 14.3]
Statistical Analysis 1: Comparison: Healthy Breastfeeding Women vs Women With IBD; This is to confirm that there is no difference in the second sampling time points in the mid-lactation period between the groups; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparison
Statistical Analysis 2: Comparison: Healthy Breastfeeding Women vs IBD Subgroup "On TNFmAb Treatment" vs IBD Subgroup "Off TNFmAb Treatment"; Test type: Superiority; p = 0.51, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 18 months from the delivery for both the mothers and infants.
Description: This is an observational study of breastfeeding women with or without IBD. Some of women with IBD are receiving treatment using monoclonal antibody against TNF (TNFmAb), which is widely known as little to no excretion into milk and is considered no risk to breastfed infants. In addition, there was no study intervention for the purpose of treatment.
Arm/Group | Women With IBD | Healthy Breastfeeding Women
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/33
Other Adverse Events (participants affected / at risk) | 0/46 | 0/33

LIMITATIONS AND CAVEATS:
This observational cohort study continued throughout the pandemic restrictions in person-to-person contact. This posed significant challenges to us. Despite this, the participating mother-infant pairs volunteered for the study. This may be the reason why many women in our IBD cohort were in remission, and those women on a severe end of IBD spectrum were not represented by our cohort, limiting the generalizability of our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03397108/Prot_SAP_ICF_000.pdf